CLINICAL TRIAL: NCT06484010
Title: Effectiveness of the Implementation of SNAPPS in Family Medicine Residency Program in Erbil: A Randomized Controlled Trial
Brief Title: Effectiveness of SNAPPS in Family Medicine Residency Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Collaborators: Arab Board of Health Specializations, Iraq (Other)
Responsible Party: Principal Investigator, Ghaith Saad Abdulnafe Shindala, Dr, Ministry Of Health / Nineveh Health Directorate
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SNAPPS Iraq
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Medical Education
Keywords: Medical education, SNAPPS, Clinical reasoning, Iraq

STUDY DESIGN:
Intervention Model Description: Thirty Family Medicine board residents and six preceptors from the department of Community and Family Medicine/ College of Medicine/ Hawler Medical University, were chosen by the convenience method and randomly distributed into two groups; the intervention group with the SNAPPS technique (first-arm) and the control group with the traditional case presentation method (2nd-arm) using a simple random number table by Microsoft Excel program, All residents was asked to prepare and present two different cases (per resident) according to their preferences during their daily training at health centers with a total of 60 case presentations (30 presentations for each group).
  data and feedback were gathered after each presentation using validated data recording sheets.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the students (participants) and the preceptors (Outcome Assessors) in each group were unaware of the other group participants, Outcome Assessors, and the method used for case presentations.
  We ensured that by asking the participants in both groups not to discuss any information regarding the study with anyone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAPPS Group (Active Comparator): The intervention was the implementation of the SNAPPS model as a method of case presentation in out-patient settings.
  Interventions: Other: SNAPPS Model of case presentation
- Control Group (No Intervention): In the control group, as both learners and preceptors are familiar with the traditional method of case presentation, no special training was required.

INTERVENTIONS:
Other: SNAPPS Model of case presentation — The intervention was the implementation of the SNAPPS model as a method of case presentation in out-patient settings.
  All preceptors and residents in the SNAPPS group were sensitized and trained one week before the beginning of case presentations and data collection by a training session that was carried out by the authors at Brayati Primary Health Center training hall for a duration of more than two hours, the session included a preview of the traditional method, introduction to the SNAPPS method, role play and doubts clarification.
  The training materials included a presentation explaining the SNAPPS method in details with examples, instructional videos, and handouts highlighting the six steps of the SNAPPS method.
  Before the beginning of the presentation by 72 hours, there was a double check by the principal investigator with all participants regarding the method and all doubts were clarified.
  Arms: SNAPPS Group

SUMMARY:
The goal of this Randomized Controlled Trial is to assess how well SNAPPS (Summarize history and findings; Narrow differentials; Analyze differentials; Probe preceptor about uncertainties; Plan management; Select case-related issues for self-study) facilitates clinical reasoning and enhances time management in an outpatient setting as a learner-centered method of case presentation when compared to the conventional method among family medicine board residents and tutors, the main objectives of the study are:

* To assess the implementation of a new technique of teaching and case presentation in family medicine residency program.
* To understand the perception of postgraduates and tutors about this new method of case presentation.

The researchers compared the outcomes of case presentations between two groups (the SNAPPS group and the control group) using dependable variables that has been used in previous researches to assess the SNAPPS versus the traditional method of case presentation.

Participants in the SNAPPS group were introduced to the SNAPPS method by a training session, while the control group needed no intervention.

Each student had to prepare and present two cases to the assigned tutor during their routine training days.

Data were collected by the tutors during each case presentation and the participants answered survey questions regarding their opinion of the case presentation.

DETAILED DESCRIPTION:
Clinical teaching's primary objectives include evaluating students' clinical reasoning abilities, advancing, and enhancing their development, as well as giving them clinical practice and feedback potential.

Whilst trying to assist postgraduate residents in improving their clinical reasoning, medical educators experience a variety of difficulties like uncooperative patients, record requirements, increasing tasks, time restraints, and productivity objectives that conflict with teaching time.

Students rarely convey their clinical reasoning or case-based doubts during traditional case presentations to preceptors, according to studies of such presentations. Instead, they tend to emphasize mostly on factual data However, the chance to consider one's own method of clinical thinking is seen as one of the most valuable components of the educational experience by both students and preceptors. Irby and Wilkerson have recently argued that there is a need for the development of time-effective teaching techniques in the clinical setting that give insights into the students' clinical reasoning strategies and doubts while also enabling the preceptor to stay completely involved in the priority areas of patient care.

Yonke and Foley questioned whether successful educational methods in the hospital setting would translate well to the office as medical education stepped from the inpatient to the outpatient setting.

Two models for enhancing clinical thinking ability-one-minute preceptor (OMP) and SNAPPS (Summarize history and findings; Narrow differentials; Analyze differentials; Probe preceptor about uncertainties; Plan management; Select case-related issues for self-study), have been well studied in the outpatient settings.

Additionally, by using these teaching models, preceptors can give trainees a more specific education without losing more precious time.

In the SNAPPS paradigm, the student presents a case to the preceptor by giving an informative summary of the pertinent information, which is followed by five steps that advocate for the expression of thinking and reasoning aloud. These actions are inspired in part by the rating scales for cognitive activity created by Connell et al.

The SNAPPS paradigm relies on a learner-teacher continuum which in the end, should be led by the learner, but may initially require coaching from the preceptor to assist the learner become comfortable and proficient with the processes. It is now both the trainer's and trainee's responsibility to ensure the prosperity of the learning process rather than just one of them.

To improve medical education in Family Medicine and other fields as well, we must comprehend and keep up with contemporary methodologies as they evolve in education.

The Aim of the study is to assess how well SNAPPS facilitates clinical reasoning and enhances time management in an outpatient setting when compared to conventional method of case presentation.

ELIGIBILITY:
Inclusion Criteria:

Residents:

* Postgraduate students.
* Pursuing the board degree in Family Medicine after completion of their M.B.Ch.B and internship.

  (16 residents from the Arabic Board of Health Specialties fellowship and 14 residents from Kurdistan Board of Medical Specialties).

Preceptors

* Tutors who worked at the department of Community and Family Medicine/ College of Medicine / Hawler Medical University.
* Frequently instructed undergraduate and postgraduate students in the family medicine teaching health facilities.

(two assistant professors and four lecturers).

Exclusion Criteria:

Family Medicine residents, who are not enrolled in the Board study (not a postgraduate student)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Total presentation length (Time in Minutes) | Data (Time) was recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The total case presentation time was measured in minutes. The comparison was made between the 2 groups' presentations depending on the mean of the total presentation time in each group.
Duration of summary (Time in Minutes) | Data (Time) was recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The duration of summary time was measured in minutes. The comparison was made between the 2 groups' presentations depending on the mean duration of summary in each group.
Number of basic clinical attributes covered | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The number of basic clinical attributes covered during each presentation was recorded and the comparison made between the two groups on the mean number of basic clinical attributed covered in each group.
Number of diagnoses kept (Dx) in differential diagnosis (DDx) | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The comparison made between the two groups on the mean number of diagnoses kept (Dx) in differential diagnosis (DDx) in each group.
Number of basic attributes in support of Diagnoses (Dx) in the differential diagnosis (DDx) | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The comparison made between the two groups on the mean number of basic attributes in support of Dx in the DDx in each group.
Number of justified diagnoses (Dx) in the differential diagnosis (DDx) | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The comparison made between the two groups on the mean number of justified diagnoses (Dx) in the differential diagnosis (DDx) in each group.
Number of distinct comparisons made between two diseases | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The comparison made between the two groups on the mean number of distinct comparisons made between two diseases in each group.
Does the student seek clarification and information by asking questions and acknowledging their uncertainties? | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The answer was Yes or No. The comparison made between the two groups depending on the percentage of those who got (Yes) or (No) in each group.
Number of uncertainties expressed and obtained clarifications | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The comparison made depending on the mean number of uncertainties expressed and obtained clarifications in each group.
Did the student discuss patient management plan? | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The answer was Yes or No. The comparison made between the two groups depending on the percentage of those who got (Yes) or (No) in each group.
Did the student Discuss case related topics and resources? | Data were recorded by the preceptors during each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The answer was Yes or No. The comparison made between the two groups depending on the percentage of those who got (Yes) or (No) in each group.

SECONDARY OUTCOMES:
Residents' Feedback on each presentation | Data were recorded by each resident after each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  Measures the residents' agreement on Likert Scale-based questionnaire (a scale used to represent people's attitudes, opinion or perception to a topic) regarding their experience in each case presentation, the format of the scale was composed of 5 level Likert items (5 indicating strongly agree whereas 1 indicating strongly disagree)
  1. Strongly disagree (minimum)
  2. Disagree
  3. Neither agree nor disagree (neutral)
  4. Agree
  5. Strongly agree (maximum)
  The Feedback of the residents in both groups was compared to each other depending on the mean of their scores.
Preceptors' Feedback on each presentation | Data were recorded by the preceptors after each case presentation, then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  Measures the preceptors' agreement on Likert Scale-based questionnaire (a scale used to represent people's attitudes, opinion or perception to a topic) regarding their experience in each case presentation, the format of the scale was composed of 5 level Likert items (5 indicating strongly agree whereas 1 indicating strongly disagree)
  1. Strongly disagree (minimum)
  2. Disagree
  3. Neither agree nor disagree (neutral)
  4. Agree
  5. Strongly agree (maximum)
  The Feedback of the preceptors in both groups was compared to each other depending on the mean of their scores.

OTHER OUTCOMES:
Diagnostic Thinking Inventory (DTI) scores | Data were recorded by each resident after the 2nd case presentation (final presentation for each resident), then analyzed using the Statistical Package for Social Sciences (SPSS, version 26) 2 weeks after all the presentations were finished.
  The Diagnostic Thinking Inventory (DTI) is a self-report instrument that has been validated to assess clinical reasoning.
  This inventory contains 41 items concerning the diagnostic thinking. Each item contains a stem, two accompanying statements and a rating scale. The scale refers to a continuum between the two statements.
  The score of each student is calculated by the summation of the rating scale score (from 1 to 6).
  The DTI questionnaire was given to the students in both groups following the final case presentation and the scores were calculated according to the DTI categories of thinking flexibility and the structure of memory.
  The randomized groups of Family Medicine residents were compared on the mean of the scores they obtained after their presentations.

CONTACTS AND LOCATIONS:
Overall Officials: Ghaith S Shindala, M.B.Ch.B, Principal Investigator — Ninevah Health Directorate/ Ministry of Health - Iraq; Nazdar E Alkhateeb, PhD.Med.Educ, Study Director — College of Medicine/ Hawler Medical University - Iraq; Ali S Dauod, JBFM, Study Director — College of Medicine/ Hawler Medical University - Iraq
Locations (1):
- Hawler Medical University/ College of Medicine, Erbil, Iraq